CLINICAL TRIAL: NCT03264625
Title: The Effects of Oral Vitamin D Supplementation on the Prevention of Peritoneal Dialysis-related Peritonitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Dong Jie, Director of PD center, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vitamin D, RCT
Record Dates: First submitted 2016-10-10; First posted 2017-08-29 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Peritoneal Dialysis-associated Peritonitis; Vitamin D Deficiency
Keywords: Cholecalciferol; Peritoneal dialysis; Peritonitis
MeSH Terms: conditions — Vitamin D Deficiency; Peritonitis | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Patients will receive oral Cholecalciferol (2000IU qd) apart from routine therapy for PD
  Interventions: Drug: Cholecalciferol (2000iu qd); Other: Routine therapy for PD
- Control group (Placebo Comparator): Patients randomized to the placebo group will receive routine therapy for PD.
  Interventions: Other: Routine therapy for PD

INTERVENTIONS:
Drug: Cholecalciferol (2000iu qd) — Patients will receive oral Cholecalciferol (2000IU qd) apart from routine therapy for PD
  Other Names: Natural Vitamin D3
  Arms: Treatment group
Other: Routine therapy for PD — Patients randomized to the placebo group will receive routine therapy for PD.

SUMMARY:
This is a pilot randomized, controlled trial of Vitamin D supplementation in patients on peritoneal dialysis to determine the feasibility of a future full-scale RCT exploring if oral administration of vitamin D3 could reduce the risk of subsequent Peritoneal dialysis-related (PD-related) peritonitis.

Aims of the study:

Aim 1: To determine the feasibility of oral vitamin D supplementation among PD patients who have recovered from a recent episode of peritonitis.

Aim 2: To examine the effect of vitamin D supplementation on the risk for peritonitis among patients on peritoneal dialysis.

DETAILED DESCRIPTION:
Patients will be screened for eligibility one month after the onset of PD-related peritonitis, those who meet the inclusion criteria will be enrolled in this study.

All consenting participants will be randomized into the vitamin D treatment group or the control group, general information and baseline biochemistry data would be collected. Patients in the treatment group will be treated with oral Cholecalciferol (2000IU/day) apart from routine treatment for PD. Those in the control group will receive routine treatment for PD. Both groups will be followed for 12 months. During the observational period, any onset of subsequent peritonitis will be recorded, serum 25(OH)D, biochemical indices will be measured every 3 months. Follow up would take place frequently, any outcome events would be recorded.

Aims and hypotheses:

Aim 1: To determine the feasibility of oral vitamin D supplementation among PD patients who have recovered from a recent episode of peritonitis.

Hypothesis1: A large、full-scale randomized controlled trail on the effects of oral vitamin D on the risk for peritonitis among PD patients is feasible.

Aim 2: To examine the effect of vitamin D supplementation on the risk for peritonitis among patients on peritoneal dialysis.

Hypothesis 2: Oral supplementation of vitamin D will reduce the risk of subsequent peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Medically stable and receiving peritoneal dialysis (PD) for>1 months
2. Age at least 18 years.
3. Serum 25(OH)D<75nmol/l (30ng/ml)
4. Adequate dialysis on evaluation, weekly Kt/V ≥ 1.5 and no clinical uremic symptoms

Exclusion Criteria:

1. Receive Vitamin D2/D3 or drugs known to alter serum 25-hydroxyvitamin D (25(OH)D) levels during the previous 12 months;
2. History of allergic reaction to Cholecalciferol;
3. Current or past malignant disease, active hepatitis or hepatic failure, acute systemic infection, active autoimmune diseases, severe digestive malabsorption or eating disorder, HIV/AIDS;
4. A high probability (assessed by the recruiting physician) of receiving a kidney transplant or transferring to hemodialysis (HD) or drop-out due to socioeconomic causes within 6 months;
5. Pregnant or breastfeeding;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2021-05-28 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate of the trial | From date of randomization until 1 year after the randomization of last participant.
  Recruitment rate of patients screened for the trial measured by percentage.
Retention rate of the trial | From date of randomization until 1 year after the randomization of last participant
  Retention rate of included patients in the trial measured by percentage.
Adherence rate of the trial | From date of randomization until 1 year after the randomization of last participant.
  Percentage of participants adherent to the dosing regimen of vitamin D in the trial.
Incidence of adverse events | From date of randomization until 1 year after the randomization of last participant.
  Incidence of adverse events measured by number of events per patient-month
Change in serum 25(OH)D level | From date of randomization until 1 year after the randomization of last participant
  Change in serum 25(OH)D level between baseline and 12 months measured by ng/ml.

SECONDARY OUTCOMES:
Difference in risk of a subsequent peritonitis measured by Hazard Ratio. | From date of randomization until the date of subsequent peritonitis, assessed up to 1 year.
  Risk of a subsequent peritoneal dialysis related peritonitis in the interventional group compared with the control group measured by Hazard Ratio.
Probability of participants who recovered after subsequent peritoneal dialysis related peritonitis. | From date of randomization until the date of documented death, assessed up to 1 year.
  Probability of participants who recovered after peritoneal dialysis-related peritonitis measured by percentage.
Risk of participants who died because of subsequent peritoneal dialysis related peritonitis. | From date of randomization until the date of documented death, assessed up to 1 year.
  Risk of participants who died because of peritoneal dialysis-related peritonitis measured by percentage.
Risk of participants who are transitioned to hemodialysis because of subsequent peritoneal dialysis related peritonitis. | From date of randomization until the date of documented transition to hemodialysis because of peritoneal dialysis related peritonitis, assessed up to 1 year.
  Risk of patients who are transferred to hemodialysis because of peritoneal dialysis related peritonitis measured by percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Dong, Study Director — Peking Universiy First Hospital
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pi HC, Ren YP, Wang Q, Xu R, Dong J. Serum 25-Hydroxyvitamin D Level Could Predict the Risk for Peritoneal Dialysis-Associated Peritonitis. Perit Dial Int. 2015 Dec;35(7):729-35. doi: 10.3747/pdi.2014.00177. Epub 2015 Jul 29. PMID 26224791
- [Background] Armas LA, Andukuri R, Barger-Lux J, Heaney RP, Lund R. 25-Hydroxyvitamin D response to cholecalciferol supplementation in hemodialysis. Clin J Am Soc Nephrol. 2012 Sep;7(9):1428-34. doi: 10.2215/CJN.12761211. Epub 2012 Jul 12. PMID 22798536
- [Derived] Zhang YH, Xu X, Pi HC, Yang ZK, Johnson DW, Dong J. The effects of oral vitamin D supplementation on the prevention of peritoneal dialysis-related peritonitis: study protocol for a randomized controlled clinical trial. Trials. 2019 Nov 28;20(1):657. doi: 10.1186/s13063-019-3784-7. PMID 31779675

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT03264625/Prot_SAP_000.pdf